CLINICAL TRIAL: NCT05983978
Title: No-biopsy Approach for the Diagnosis of Celiac Disease: Definition of Cut-off Points for Different IgA Anti-tissue Transglutaminase Assays
Brief Title: No-biopsy Approach in Celiac Disease: Cut-off Points for IgA Anti-tissue Transglutaminase Assays
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Hospital Universitari Mutua Terrassa (Unknown); Hospital Sant Joan de Deu (Other); Hospital Universitario Ramon y Cajal (Other); Hospital Universitario Lucus Augusti (Other); Hospital Universitario Fundación Jiménez Díaz (Other); Instituto de Investigación Sanitaria Hospital Clínico San Carlos (Unknown)
Responsible Party: Principal Investigator, Marta Molero, Doctor, Instituto de Investigación Hospital Universitario La Paz
Other Study IDs: PI-5473
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Celiac Disease
Keywords: anti-transglutaminase IgA; no-biopsy approach
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The main objective of this multicenter and observational study is to define the optimal threshold of different commercially available IgA anti-transglutaminase (tTG-IgA) antibody assays for celiac disease diagnosis (CD) avoiding the need for an intestinal biopsy.

The main questions to be answered are:

* Is the anti-tTG-IgA titer cut-off above 10 times the upper limit of normal (ULN) useful in all anti-tTG IgA assays?
* Is the diagnostic performance of the newly defined cut-offs of anti-tTG-IgA the same in all the evaluated assays?
* Is the dynamic of the anti-tTG-IgA levels after the introduction of the gluten-free diet (GFD) similar across the different assays included in the study?

This is a prospective multicenter study that will enroll pediatric and adult patients with new-onset CD during the years 2023 and 2024. Serum from these patients will be collected for the determination of anti-tTG-IgA according to the local methodology (participating hospital) and by the anti-tTG IgA assays most commonly used in our country, which will be centralized in the same reference center (Hospital Universitario La Paz).

ELIGIBILITY:
Inclusion criteria:

* Patients, on gluten-containing diet, with TGt-IgA antibodies > Upper Limit of Normal (ULN) and intestinal biopsy confirming celiac disease (CD).
* Patients with TCRγδ+ >10% combined with decrease NK-like intraepithelial lymphocytes in the intestinal epithelium.
* Paediatric patients who meet ESPGHAN criteria (TGt-IgA antibodies >10xULN) without duodenal biopsy performed.

Exclusion criteria:

* Patients already diagnosed with CD.
* Patients who refused duodenal biopsy.
* Patients with primary or secondary immunodeficiencies.
* Patients with malignancy.
* Recruited patients whose remaining serum cannot be sent to the reference centre, whose biopsies are of poor quality or who nod not sign the informed consent from.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be consecutively recruited from the gastroenterology departments (either adult or pediatric) of the participating hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Anti-transglutaminase-IgA titer | The tTG-IgA will be measured at the time of patient recruitment and at the first follow-up (3-6 months from the start of the gluten-free diet).
  To define the optimal threshold for anti tTG-IgA levels using different commercially available assays that provide a positive predictive value of 100%.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Molero-Luis, Dr, Principal Investigator — Hospital Universitario La Paz
Locations (6):
- Spain (6):
  - Hospital Mutua Terrassa, Terrassa, Barcelona
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Sant Joan de Deu, Barcelona
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario Fundación Jimenez Diaz, Madrid